CLINICAL TRIAL: NCT00106483
Title: Autoimmunity and Coronary Artery Disease - Ancillary to CARDIA
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Darcy Majka, Assistant Professor in Medicine & Preventive Medicine, Northwestern University
Other Study IDs: 1291; R21HL079057 (NIH)
Record Dates: First submitted 2005-03-24; First posted 2005-03-25 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases
Keywords: Cardiovascular Diseases; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Coronary Artery Risk Development in Young Adults: There were no interventions.

SUMMARY:
To test the primary hypothesis that individuals with pre-clinical connective tissue disease related autoimmunity are more likely to demonstrate subsequent development of sub-clinical coronary artery disease.

DETAILED DESCRIPTION:
BACKGROUND:

Connective tissue diseases have been identified as risk factors for coronary artery disease (CAD). Patients with connective tissue diseases such as rheumatoid arthritis and systemic lupus erythematosus have a high prevalence of CAD and are younger than expected at the onset of CAD. It has been proposed that the association between these connective tissue diseases and CAD is related to inflammation. Furthermore, circulating autoantibodies have been identified in CAD and it has been hypothesized that CAD may have autoimmune features. Circulating autoantibodies exist prior to connective tissue disease development and the presence of such autoantibodies in asymptomatic individuals is a predictor of future clinical connective tissue disease. Although the association between connective tissue disease and CAD has been established, an association between pre-clinical circulating autoantibodies and early CAD has not yet been explored.

DESIGN NARRATIVE:

To test this hypothesis, the following specific aims are proposed using the CARDIA database: 1) Determine the association between autoimmunity measured in stored sera collected in 1992 and the subsequent development of sub-clinical CAD measured in 2000 and 2005. 2) Assess whether autoimmunity measured in 1992 predicts future increased levels of C-reactive protein (CRP) and whether the relationship between autoimmunity and CAD is mediated by CRP level. These aims will be accomplished by a team of investigators within the Division of Rheumatology and Department of Preventive Medicine at Northwestern University. The CARDIA database is a product of the Coronary Artery Risk Development in Young Adults (CARDIA) study, a prospective cohort of 5108 subjects followed since 1985 for development of novel cardiac risk factors. With its extensive epidemiologic database and stored serum collected serially and available from 3500 individuals over the past 20 years, the CARDIA study is an ideal resource for this study.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All CARDIA participants with serum available in 1992 and coronary calcification measure in years 2000 and 2005.
Sampling Method: Non-Probability Sample
Enrollment: 3020 (Actual)
Dates: Start 2005-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Coronary artery calcification (CAC) | 8 years
  serum samples already collected by they CARDIA study in 1992 were tested by our ancillary study for autoantibodies and we analyzed whether autoantibody positivity was associated with CAC over 13 years of follow up in the CARDIA study. CAC was measured by the CARDIA study in 2000 and 2005.

CONTACTS AND LOCATIONS:
Overall Officials: Darcy Majka, MD MS, Principal Investigator — Northwestern University School of Medicine